CLINICAL TRIAL: NCT01476436
Title: Low Carbohydrate Diet - Effect on Plasma Lipids and Metabolic Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Kjetil Retterstøl, Associate professor, MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: REK195276
Record Dates: First submitted 2011-08-11; First posted 2011-11-22 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Overweight and Obesity; Type IIb Hyperlipidaemia; Hypercholesterolemia Aggravated
Keywords: Cardio vascular risk factors
MeSH Terms: conditions — Overweight; Obesity; Hyperlipoproteinemia Type II | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCHF diet (Experimental): Advice of a diet low in carbohydrate
  Interventions: Other: Low carbohydrate dietary advice; Other: Continue usual diet
- Usual diet (Active Comparator): Subjects shall continue to eat their usual daily diet with no low carbohydrate intervention
  Interventions: Other: Continue usual diet

INTERVENTIONS:
Other: Low carbohydrate dietary advice — Dietary advice
  Other Names: Dietary advice
  Arms: LCHF diet
Other: Continue usual diet — Dietary advice
  Other Names: Lifestyle counseling to continue usual diet

SUMMARY:
Low carbohydrate diet may influence the plasma lipid levels.

DETAILED DESCRIPTION:
Fasting plasma lipids will be measured in healthy volunteer randomized to low carbohydrate diet or usual diet for a period

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion criteria:

Any disease or use of prescriptional medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Percent change in mean LDL-cholesterol after intervention with low carbohydrate diet | From baseline to study end

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Retterstøl, MD PhD, Principal Investigator — University of Oslo, Faculty of Medicine, Institute of Basic Medical Sciences, Department of Nutrition
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Homepage — http://www.med.uio.no/imb/english/